CLINICAL TRIAL: NCT02289352
Title: A Randomized, Double-Blind, Multiple-Site, Placebo-Controlled, Parallel-Design Study to Evaluate the Safety and Therapeutic Equivalence of Brimonidine Topical Gel, 0.33% (Watson Laboratories, Inc., USA) to Reference Product Mirvaso® (Brimonidine) Topical Gel, 0.33% (Galderma Laboratories, L.P., USA) in Patients With Moderate to Severe Facial Erythema Associated With Rosacea
Brief Title: Randomized, Double-blind, Multiple-site, Placebo-controlled, Parallel-design Study in Patients With Moderate to Severe Facial Erythema Associated With Rosacea
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Actavis Inc. (Industry)
Collaborators: Watson Laboratories, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 71304906
Record Dates: First submitted 2014-10-31; First posted 2014-11-13 (Estimated); Results first posted 2020-01-14 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Rosacea
MeSH Terms: conditions — Rosacea | interventions — Brimonidine Tartrate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- brimonidine 0.33% gel (Experimental): Brimonidine Topical Gel, 0.33%, 30 gram fill (Watson Laboratories, Inc., USA)
  Interventions: Drug: Brimonidine
- Mirvaso gel (Active Comparator): Mirvaso® (brimonidine) topical gel, 0.33% (Galderma Laboratories, L.P., USA)
  Interventions: Drug: Brimonidine
- Placebo (Placebo Comparator): Topical gel base only (Watson Laboratories Inc., USA)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Brimonidine
  Arms: Mirvaso gel; brimonidine 0.33% gel
Drug: placebo
  Arms: Placebo

SUMMARY:
A Randomized, Double-Blind, Multiple-Site, Placebo-Controlled, Parallel-Design Study to Evaluate the Safety and Therapeutic Equivalence of Brimonidine Topical Gel, 0.33% (Watson Laboratories, Inc., USA) to Reference Product Mirvaso® (brimonidine) topical gel, 0.33% (Galderma Laboratories, L.P., USA) in Patients with Moderate to Severe Facial Erythema Associated with Rosacea

DETAILED DESCRIPTION:
Up to 462 patients 18 years of age and older, with confirmed clinical diagnosis of rosacea will be enrolled to have 413 in the modified intent-to-treat (mITT) population and 371 in the per-protocol (PP) population. Patients should have fewer than 3 facial inflammatory lesions, and moderate to severe erythema according to both Clinician's Erythema Assessment (CEA) and Patient's Self-Assessment (PSA).

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant, non-lactating female, 18 years of age or older.
2. Signed informed consent form, which meets all criteria of current FDA regulations.
3. Females of child bearing potential must not be pregnant or lactating at Screening and Randomization (as confirmed by a negative urine pregnancy test with a sensitivity of less than 25 mlU/mL or equivalent units of human chorionic gonadotropin). Women of childbearing potential must agree to the use of a reliable method of contraception (e.g., total abstinence, IUD, a double-barrier method [such as condom plus diaphragm with spermicide], oral, transdermal, injected or implanted non- or hormonal contraceptive), throughout the study. A sterile sexual partner is not considered an adequate form of birth control.

   All females will be considered to be of childbearing potential unless they:
   * Are post-menopausal, defined as women who have been amenorrheic for at least 12 consecutive months, without other known or suspected primary cause.
   * Have been sterilized surgically or who are otherwise proven sterile (i.e., total hysterectomy, or bilateral oophorectomy) with surgery at least 4 weeks prior to Screening. Tubal ligation will not be considered a surgically sterile method.

   Female patients of childbearing potential are defined as:
   * Women without prior hysterectomy, or who have had any evidence of menses in the past 12 months.
   * Females who have been amenorrhea for ≥ 12 months, but the amenorrhea is possibly due to other causes, including prior chemotherapy, anti-estrogens, or ovarian suppression.
4. Have a clinical diagnosis of facial rosacea and fewer than 3 inflammatory lesions on the face at Screening and at Randomization (before drug application on Day 1).
5. Have moderate to severe facial erythema according to both CEA and PSA (i.e., an erythema score of 3 or more for each of the CEA and PSA) at Screening and at Randomization (before drug application on Day 1).
6. Free from any systemic or dermatologic disorder (other than rosacea) that, in the opinion of the Investigator, will interfere with the study evaluations or increase the risk of AEs.
7. Willing to minimize external factors that might trigger rosacea flare-ups (e.g., hot environments, prolonged sun exposure, strong winds and emotional stress) within 24 hours of the Screening and Randomization visit.
8. Any skin type or race, providing the skin pigmentation will allow discernment of erythema.
9. Willingness and capability to cooperate to the extent and degree required by the protocol.

Exclusion Criteria:

1. Patients with particular forms of rosacea (rosacea conglobata, rosacea fulminans, isolated rhinophyma, isolated pustulosis of the chin) or other concomitant facial dermatoses similar to rosacea, such as peri-oral dermatitis, demodicidosis, facial keratosis pilaris, seborrheic dermatitis, acute lupus erythematosus, or actinic telangiectasia, that are present on the face (i.e., 5 areas: chin, nose, both cheeks, and forehead), that in the opinion of the Investigator would interfere with study evaluations.
2. Have 3 or more facial inflammatory lesions of rosacea.
3. Have an erythema score of 2 (mild), 1 (almost clear), or 0 (clear) on the CEA and/or the PSA at Screening and at Randomization (before drug application on Day 1).
4. Patients with excessive facial hair (beards, sideburns, mustaches, etc.) that would interfere with the diagnosis or assessment of rosacea.
5. Patients with moderate to severe telangiectasial masses in the 5 areas of the entire face: forehead, chin, nose and each cheek, that would interfere with study evaluations.
6. History of hypersensitivity or allergy to Mirvaso® including the active ingredient brimonidine tartarate or other component within the formulation.
7. Facial laser surgery for telangiectasia (or other conditions) within 6 weeks prior to randomization.
8. Exposed to excessive ultraviolet (UV) radiation within 1 week before screening or randomization visit and/or patient was unwilling to refrain from excessive exposure to UV radiation during the course of the study.
9. History of blood dyscrasia.
10. Current diagnosis of Raynaud's syndrome, thromboangiitis obliterans, orthostatic hypotension, severe cardiovascular disease, cerebral or coronary insufficiency, renal or hepatic impairment, scleroderma, Sjögren's syndrome, or depression, or any other condition causing uncontrolled blood flow or blood pressure.
11. Females who are pregnant, lactating or likely to become pregnant during the study.
12. Significant history or current evidence of chronic infectious disease, system disorder, organ disorder or other medical condition that in the Investigator's opinion would place the study patient at undue risk by participation.
13. Patients with severe, unstable or uncontrolled cardiovascular disease.
14. Patients who meet study restrictions at Screening and Randomization and/or unwillingness to comply with all restricted treatments
15. Receipt of any drug as part of a research study within 30 days before dosing.
16. Employees of the research center or Investigator.
17. Previous participation in this study.
18. Patients who are unable and/or unwilling to follow the study requirements, and procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 462 (Actual)
Dates: Start 2014-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nageshwar R Thudi, Ph.D., Study Director — Actavis Inc.
Locations (16):
- United States (16):
  - Investigator site 2, Hot Springs, Arkansas
  - Investigator site 16, Long Beach, California
  - Investigator site 5, Miami, Florida
  - Investigator site 7, Miami, Florida
  - Investigator site 8, Miramar, Florida
  - Investigator site 6, Ormond Beach, Florida
  - Investigator site 3, Carmel, Indiana
  - Investigator site 9, Louisville, Kentucky
  - Investigator site 14, Fridley, Minnesota
  - Investigator site 15, Henderson, Nevada
  - Investigator site 1, Albuquerque, New Mexico
  - Investigator site 10, High Point, North Carolina
  - Investigator site 11, Beachwood, Ohio
  - Investigator site 4, Nashville, Tennessee
  - Investigator site 13, College Station, Texas
  - Investigator site 12, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 514 patients were screened for study participation and 462 patients were randomized and included in the statistical analysis.
  The populations for this study included the Safety population, the Per-Protocol (PP) population and the modified Intent-to-Treat (mITT) Population.
Groups:
- Test: Brimonidine 0.33% Gel: Brimonidine Topical Gel, 0.33%, 30 gram fill (Watson Laboratories, Inc., USA)
  Participants applies a once-daily application of brimonidine gel (pea-sized amount to each of 5 areas of the entire face for 7 days).
- Reference: Mirvaso 0.33% Gel: Mirvaso® (brimonidine) topical gel, 0.33% (Galderma Laboratories, L.P., USA)
  Participants applies a once-daily application of brimonidine gel (pea-sized amount to each of 5 areas of the entire face for 7 days).
- Placebo Gel Vehicle: Topical gel base only (Watson Laboratories Inc., USA)
  Participants applies a once-daily application of brimonidine gel (pea-sized amount to each of 5 areas of the entire face for 7 days).
Period: Overall Study
Arm/Group | Test: Brimonidine 0.33% Gel | Reference: Mirvaso 0.33% Gel | Placebo Gel Vehicle
Started | 199 | 199 | 64
Safety Population (Randomized participants who received the study drug.) | 199 | 199 | 64
mITT Population (Randomized participants, at least one dose, pre and post assessments during at least one visit (2/3)) | 191 | 193 | 58
PP Population (Participants completed all visits and assessments, dose compliance, and followed restrictions.) | 173 | 173 | 54
Completed | 198 | 198 | 64
Not Completed | 1 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Test:Brimonidine 0.33% Gel; Reference: Mirvaso 0.33% Gel; Placebo Gel Vehicle: Participants applies a once-daily application of brimonidine gel (pea-sized amount to each of 5 areas of the entire face for 7 days).
- Total: Total of all reporting groups
Arm/Group | Test:Brimonidine 0.33% Gel | Reference: Mirvaso 0.33% Gel | Placebo Gel Vehicle | Total
Number analyzed (Participants) | 199 | 199 | 64 | 462
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 163 | 167 | 54 | 384
  >=65 years | 36 | 32 | 10 | 78
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 151 | 156 | 53 | 360
  Male | 48 | 43 | 11 | 102
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 60 | 65 | 19 | 144
  Not Hispanic or Latino | 139 | 134 | 45 | 318
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 198 | 198 | 64 | 460
  More than one race | 1 | 1 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Primary: Percentage of Treatment Success on Day 7
Description: Percentage of patients with a clinical response of treatment success on Day 7 (± 1). Treatment success is defined as at least a 2-grade improvement on both CEA and PSA scores from baseline (pre-dose) on Day 7 (± 1) to 6 hours post-application on Day 7 (± 1).
Time Frame: 7 days
Population: Participants in the mITT Population that were evaluated for percentage of treatment successes.
Measure: Number; unit: percentage of participants
Groups:
- Test: Brimonidine 0.33% Gel: Brimonidine Topical Gel, 0.33%, 30 gram fill (Watson Laboratories, Inc., USA)
  Test Brimonidine
- Reference: Mirvaso 0.33% Gel: Mirvaso® (brimonidine) topical gel, 0.33% (Galderma Laboratories, L.P., USA)
  Reference Brimonidine
- Placebo: Vehicle gel
Arm/Group | Test: Brimonidine 0.33% Gel | Reference: Mirvaso 0.33% Gel | Placebo
Number analyzed (Participants) | 191 | 193 | 58
percentage of participants | 9.95 | 10.36 | 0
Statistical Analysis 1: Comparison: Test: Brimonidine 0.33% Gel vs Reference: Mirvaso 0.33% Gel; Test type: Equivalence — If the 90% confidence interval for the absolute difference between the proportion of patients considered a treatment success (at least a 2-grade improvement on both CEA and PSA over 6 hours+/-10 minutes) in the Test and Reference groups is contained within the range [-20%, +20%], then bioequivalence of the Test product to the Reference product is considered to have been demonstrated; Mean Difference (Net) = -0.58, 90% CI 2-sided [-6.49 to 5.33]
Statistical Analysis 2: Comparison: Test: Brimonidine 0.33% Gel vs Placebo; Test type: Superiority; p < 0.0001, t-test, 2 sided
Statistical Analysis 3: Comparison: Reference: Mirvaso 0.33% Gel vs Placebo; Test type: Superiority; p < 0.0001, t-test, 2 sided

2. Secondary Outcome: Percentage of Patients With a Clinical Response of Treatment Success on Day 1
Time Frame: 1 day
Measure: Number; unit: percentage of participants
Groups:
- Placebo: Placebo Vehicle gel
Arm/Group | Test: Brimonidine 0.33% Gel | Reference: Mirvaso 0.33% Gel | Placebo
Number analyzed (Participants) | 191 | 193 | 58
percentage of participants | 30.89 | 30.89 | 8.62
Statistical Analysis 1: Comparison: Test: Brimonidine 0.33% Gel vs Reference: Mirvaso 0.33% Gel; Test type: Equivalence — The secondary efficacy variable is the proportion of patients with a clinical response of treatment success on Day 1. If the 90% confidence interval for the absolute difference between the proportion of patients considered a treatment success (at least a 2-grade improvement on both the CEA and PSA over 6 hours+/-10 minutes) in the Test and Reference groups is contained within the range [-20%, 20%], then bioequivalence of the Test to Reference product is considered to have been demonstrated; Mean Difference (Net) = 6.94, 90% CI 2-sided [-1.54 to 15.41]
Statistical Analysis 2: Comparison: Test: Brimonidine 0.33% Gel vs Placebo; Test type: Superiority; p < 0.0001, t-test, 2 sided
Statistical Analysis 3: Comparison: Reference: Mirvaso 0.33% Gel vs Placebo; Test type: Superiority; p = 0.0045, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Baseline to Day 7
Description: Adverse events were collected from participants who were randomized and received the study drug.
Arm/Group | Test:Brimonidine 0.33% Gel | Reference: Mirvaso 0.33% Gel | Placebo Gel Vehicle
All-Cause Mortality (participants affected / at risk) | 26/199 | 22/199 | 4/64
Serious Adverse Events (participants affected / at risk) | 0/199 | 0/199 | 0/64
Other Adverse Events (participants affected / at risk) | 26/199 | 22/199 | 4/64
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test:Brimonidine 0.33% Gel (N=199) | Reference: Mirvaso 0.33% Gel (N=199) | Placebo Gel Vehicle (N=64)
Dry Mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Application site acne (General disorders) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Heart Rate Increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Burning sensation (Nervous system disorders) | 4 (4) | 9 (10) | 0 (0)
Stress (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 6 (11) | 5 (8) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Application site erythema (General disorders) | 5 (13) | 7 (11) | 0 (0)
Application site irritation (General disorders) | 1 (1) | 0 (0) | 0 (0)
Application site pain (General disorders) | 5 (5) | 2 (2) | 0 (0)
Application site papules (General disorders) | 1 (1) | 0 (0) | 0 (0)
Application site pruritus (General disorders) | 4 (4) | 2 (3) | 1 (1)
Application site warmth (General disorders) | 2 (10) | 2 (4) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 4 (4) | 6 (7) | 0 (0)
Hyperaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results of the study may be published or presented by the Investigator(s) after the review by, and in consultation and agreement with the Sponsor, and such that confidential or proprietary information is not disclosed.